CLINICAL TRIAL: NCT00708825
Title: Reverse-Loop Upper Arm Arteriovenous Graft for Chronic Hemodialysis
Brief Title: Reverse-Loop Upper Arm Arteriovenous Graft
Status: Suspended | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Min-Sheng General Hospital (Other)
Responsible Party: Chih-Yang Chan, MD, PhD, Far Eastern Memorial Hospital
Other Study IDs: FEMH 97018
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Blood Vessel Prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — prosthetic vascular graft (ePTFE)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: surgical outcome, observation

SUMMARY:
Background: A conventional configured prosthetic arteriovenous graft (AVG) usually wastes most upper arm vessels that a reverse-loop design may conserve. This study examined the feasibility of the AVG construction and its outcome.

Methods: Retrospective review of clinical outcomes of reverse-loop upper arm AVG patients. Measures included hemodialysis function, duplex scan, procedural complications, and follow-up interventions

ELIGIBILITY:
Inclusion Criteria:

* compromized forearm and elbow options

Exclusion Criteria:

* unstable

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: uremic patient, compromized forarm and elbow options
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
functional event-free primary patency | event-free time

SECONDARY OUTCOMES:
Measures included hemodialysis function, duplex scan, procedural complications, and follow-up interventions. | events (month)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Yang Chan, MD, PhD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan